CLINICAL TRIAL: NCT06326255
Title: The Effects of Laughter Yoga on Reducing Depression and Anxiety in Children With Autism Spectrum Disorder (ASD)and Parenting Stress in Their Parents: a Pilot Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of Laughter Yoga in Children With Autism Spectrum Disorder and Their Parents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LAM Chung Yan Hemio (Other)
Responsible Party: Sponsor-Investigator, LAM Chung Yan Hemio, PhD student, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LYASD
Record Dates: First submitted 2024-03-04; First posted 2024-03-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Parenting Stress; Depression; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laughter Yoga Group (Experimental): The intervention is a laughter yoga program consisting of 12 sessions, two 1-hour sessions per month.
  Interventions: Behavioral: laughter yoga
- wait-list-control group (No Intervention): Participants will receive the same intervention after the 3-Months Follow-up (T2).

INTERVENTIONS:
Behavioral: laughter yoga — each class, including warm-up exercises, laughter yoga exercises, breathing and a relaxation session and sharing
  Arms: Laughter Yoga Group

SUMMARY:
This is a pilot randomised controlled trial to explore the acceptability and feasibility of laughter yoga about anxiety and depression reduction in children with ASD and parenting stress reduction for their parents. Hypotheses of this study include:

1. Laughter yoga is acceptable to children with ASD and their parents.
2. Laughter yoga is feasible for anxiety and depression reduction in children with ASD and parenting stress reduction in their parents.
3. Participants in the experimental group will have significantly more reduction in depression, anxiety and parental stress than those in the wait-list-control group.

DETAILED DESCRIPTION:
The intervention is a laughter yoga programme consisting of twelve sessions (biweekly). Sixty-six children with ASD and their father or mother from local autism support groups will join this study. Participants will be given an information sheet. Participants will be fully informed about laughter yoga's details, benefits and risks. All participants voluntarily take part in this study. If the family agrees to participate in this study, the parent will sign the consent form. Families will be randomized into an experimental group or a wait-list-control group. Before the laughter yoga programme, baseline data (T0) will be collected. The experimental group (n=33) will attend the twelve classes led by a certified laughter yoga trainer in an activity room that is suitable for indoor exercise. A research assistant will assist the laughter yoga teacher and provide first aid if needed. Parents will complete the questionnaire again immediately at the Programme End (T1) and at a 3-month follow-up (T2). The wait-list-control group (n=33) will receive the same laughter yoga programme after 3-month follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

THE CHILD should:

* aged 8 to 12
* be diagnosed with autism spectrum disorder (according to either The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) or International Classification of Diseases 11th), and
* able to read and understand Chinese and Cantonese, and
* have a parent (father or mother) participating in this study together.

THE PARENT should:

* be able to read and understand Chinese and Cantonese, and
* willing to attend the laughter yoga classes with their child, and
* willing to complete the required post-test.

Exclusion Criteria:

THE CHILD:

* has recently undergone surgery, or
* has a primary diagnosis not ASD, or
* has an intelligence quotient lower than 70, or
* has been diagnosed low functioning ASD, or
* has severe behavioral problems, or
* is receiving medical treatment for anxiety or depression at the start of the laughter yoga program.

THE PARENT has:

* recently undergone surgery, or
* been diagnosed with a psychiatric disorder, or
* no child with ASD is willing to participate in this study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Baseline (immediately before intervention)
  The proportion of eligible potential participants that agree to take part in.
Attrition rate | 3 Months Follow-up (9 months from baseline)
  The proportion of recruited participants that withdraw from the study at any time.
Attendance rate | Each laughter yoga session, total 12 time points
  The number and percentage of families attend each laughter yoga session.
Perception on laughter yoga | Programme end (6 months from Baseline)
  Families in the laughter yoga group will be interviewed to explore their perception of laughter yoga and its benefits.
Difficulties in laughter yoga | Programme end (6 months from Baseline)
  Families in the laughter yoga group will be interviewed to explore difficulties when they practiced laughter yoga.
Safety issues | Programme end (6 months from Baseline)
  Families in the laughter yoga group will be interviewed and explore any discomfort during or after the laughter yoga.

SECONDARY OUTCOMES:
Depression | at baseline (immediately before intervention) , Programme end (6 months from Baseline) and 3-month follow-up (9 months from Baseline)
  Parents will rate the 10 items related to their children's depression in the Revised Child Anxiety and Depression Scale - Parent Version. The scoring ranges from 0 to 30, with higher scores indicating greater severity of symptoms of depression.
Anxiety | at baseline (immediately before intervention) , Programme end (6 months from Baseline) and 3-month follow-up (9 months from Baseline)
  Parents will rate their children's social phobia (9 items, score from 0 to 27), panic disorder(9 items, score from 0 to 27), separation anxiety (7 items, score from 0 to 21), generalized anxiety (6 items, score from 0 to 18) and obsessive-compulsive behaviour (6 items, score from 0 to 18) in the Revised Child Anxiety and Depression Scale (RCADS) - Parent Version, with higher scores indicating greater severity of symptom of anxiety.
Parenting Stress | at baseline (immediately before intervention) , Programme end (6 months from Baseline) and 3-month follow-up (9 months from Baseline)
  Parents will complete the Chinese version of the Parenting Stress Index - Fourth Edition Short Form (PSI-4-SF), from 36 to 180 (36 items), with higher scores indicating a greater level of parenting stress.
Child-parent Relationships | Programme end (6 months from Baseline)
  Families in the laughter yoga group will be interviewed to assess whether any child-parent relationships have changed since practicing laughter yoga.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yan Lam, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Revised Child Anxiety and Depression Scale (RCADS) — https://www.corc.uk.net/outcome-experience-measures/revised-childrens-anxiety-and-depression-scale-rcads/
- See also: Official website of Chinese version of the Parenting Stress Index, Fourth Edition Short Form — https://www.psy.com.tw/ec99/ushop20128/goodsdescr.asp?prod_id=87470&parent_id=118&category_id=123